CLINICAL TRIAL: NCT06489327
Title: Comparing Two Doses of Oral Melatonin as Premedication in Children Undergoing Surgery: A Double-Blind Randomized Trial
Brief Title: Comparing Two Doses of Oral Melatonin as Premedication in Children Undergoing Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Al-Ayen Iraqi University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 042/2021/Babel
Record Dates: First submitted 2024-06-22; First posted 2024-07-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-07

CONDITIONS: Preoperative Anxiety
Keywords: preoperative anxiety; general anesthesia; major surgery; oral melatonin; placebo; premedication
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1st group: melatonin 0.2 mg/kg group (Active Comparator): patients will receive oral melatonin at a dose of 0.2 mg/kg
  Interventions: Drug: melatonin (Circadin ®) 0.2 mg/kg
- 2nd group: M04 groupmelatonin 0.4 mg/kg group (Active Comparator): patients will receive oral melatonin at a dose of 0.4 mg/kg
  Interventions: Drug: melatonin (Circadin ®) 0.4 mg/kg
- 3rd group: placebo group (Placebo Comparator): patients will receive oral placebo premedication
  Interventions: Drug: placebo group

INTERVENTIONS:
Drug: melatonin (Circadin ®) 0.2 mg/kg — Patients will receive oral melatonin at a dose of 0.2 mg/kg as premedication in the morning of the surgery, 90 minutes before the induction of anesthesia, with a maximum dose of melatonin set at 10 mg.
  Arms: 1st group: melatonin 0.2 mg/kg group
Drug: melatonin (Circadin ®) 0.4 mg/kg — Patients will receive oral melatonin at a dose of 0.4 mg/kg as premedication in the morning of the surgery, 90 minutes before the induction of anesthesia, with a maximum dose of melatonin set at 10 mg.
  Arms: 2nd group: M04 groupmelatonin 0.4 mg/kg group
Drug: placebo group — Patients will receive oral placebo as premedication in the morning of the surgery, 90 minutes before the induction of anesthesia, with a maximum dose of melatonin set at 10 mg.
  Arms: 3rd group: placebo group

SUMMARY:
Preoperative anxiety is a common issue in pediatric anesthesia. Children often experience anxiety and uneasiness due to uncertain outcomes. Surgery and anesthesia are among the most traumatic experiences for children, often considered anxiety-inducing medical treatments. Because they lack control over their environment and circumstances, children undergoing medical procedures typically experience significant unease or anxiety. Several studies have reported that 50%-80% of children experience preoperative anxiety.

In order to reduce kids anxiety intensity, several measures are utilized. These strategies are either pharmacological, psychological, or behavioural. Benzodiazepines are popular drugs that can reduce anxiety in children. The most used one in premedication is midazolam. It is a rapid-acting benzodiazepine that has a short elimination half-life. It has sedative, anxiolytic, hypnotic, and anterograde amnesic effects. Midazolam, on the other hand, might have a number of negative consequences, including paradoxical reactions, interactions with opioids, excessive sedation, disorientation, and reduced psychomotor performance.

Melatonin enhances anti-nociceptive effects, most prominently through the modulation of MT1/MT2 receptors in the brain and spinal cord. In addition, it has been demonstrated that melatonin can interact with additional receptors, including those in the GABAergic system, the nitric oxide (NO)arginine route, the N-Methyl-D-aspartate (NMDA) system, and the dopaminergic system, to produce anti-nociceptive and anti-allodynic effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex
* age from 4 to 14 years
* Patients with American society Anesthesiologist physical status I and II
* Patients undergoing elective surgeries

Exclusion Criteria:

* ASA more than III
* Drug allergy.
* Gastrointestinal disorders.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2026-07-12 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
preoperative anxiety | 24 hours
  The child's anxiety level will be assessed by Visual analogue scale-anxiety (VAS-A). The VAS-A consists of a 100 mm horizontal line; the left edge of the line is marked as "calm," while the other end shows "maximum anxiety." The patients were asked to assess their own anxiety and mark it on the anxiety line.

SECONDARY OUTCOMES:
preoperative sedation | 24 hours
  The sedation level will be assessed using Ramsay Sedation Scale. It divides a patient's level of sedation into six categories ranging from severe agitation at 1 to deep coma at 6.

CONTACTS AND LOCATIONS:
Overall Officials: Neveen Kohaf, ph.d, Principal Investigator — Al-Azhar University
Locations (2):
- Facualty of Pharmacy, Al Azhar University, Cairo, Cairo Governorate, Egypt
- Al-Ayen Univerisity, Madīnat Bābil, Babel, Iraq

IPD SHARING:
Plan to Share IPD: Yes
data will be shared upon resealable request from the principal investigator
Supporting Information: Study Protocol, SAP